CLINICAL TRIAL: NCT05654597
Title: French Validation of the CAPTURE Case Finding Tool for Obstructive Respiratory Disease
Status: Terminated | Type: Observational
Why Stopped: Futility analysis showed that the probability to validate out hypothesis was near from 15%
Sponsor: Groupe Hospitalier du Havre (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A00209-34
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lung Diseases; Lung Diseases, Obstructive; Obstructive Pulmonary Disease
Keywords: COPD; Asthma; Case finding
MeSH Terms: conditions — Lung Diseases; Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants aged 40 or more, without diagnosis of COPD or asthma: Men and women attending aged 40 or more, without previous diagnosis of chronic obstructive pulmonary disease or asthma.
  Interventions: Other: CAPTURE tool; Other: Spirometry

INTERVENTIONS:
Other: CAPTURE tool — CAPTURE 5-item questionnaire and a selected use of peak expiratory flow measurement.
Other: Spirometry — Spirometry performed with a portable device, used for comparison with the CAPTURE tool.

SUMMARY:
The objective of this multicentre prospective study is to validate CAPTURE as a French case finding tool for undiagnosed patients suffering from obstructive pulmonary disease.

DETAILED DESCRIPTION:
A large number of healthcare professional across the country will screen participants.

Participants willing to participate will have a short interview, and then will have to answer the 5-item CAPTURE questionnaire. They will be assisted to perform a peak expiratory flow measurement with a portable device. The comparison will be made between the CAPTURE decision and a portable spirometry assessing the presence or not of an obstructive disorder.

Patient screened either by the tool or the spirometry will be addressed to a doctor. Follow-up at 6 months will be set up in order to assess the entry or not of those patients to an approved health care pathway.

At the end of each center's participation, a questionnaire will be sent to all healthcare professionals working on the study, to assess the ease of use of spirometry and the CAPTURE tool and its possible implementation in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* People aged 40 or more,
* Provision of dated and signed informed consent form,
* Currently being treated by a healthcare professional,
* Patients affiliated to the french social security system.

Exclusion Criteria:

* Patients previously diagnosed with COPD or asthma,
* Patients with any condition making them unable to perform spirometry or answer a short questionnaire,
* Patients unable to give free and informed consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult men and women over 40 years old will be recruited from a broad range of healthcare professional in primary care across the country. Any patient attending an appointment will be screened for inclusion.
Sampling Method: Probability Sample
Enrollment: 1002 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity and area under the ROC curve of the CAPTURE tool | Baseline
  Sensitivity, specificity and area under the ROC curve of the CAPTURE tool; i.e. its ability to identify undiagnosed patients with an obstructive ventilatory disorder assessed with a portable spirometry.

SECONDARY OUTCOMES:
Number of patients who have taken steps to enter a healthcare pathway 6 months after the referral to a doctor | 6 months after
  Number of patients screened by the CAPTURE tool who have taken steps to enter a healthcare pathway 6 months after the referral to a doctor, i.e. the impact of the screening process at 6 months on patient diagnosis, management and follow-up.
Primary care investigators' opinion of the CAPTURE tool used in this study | Baseline to 2 years
  Responses on a Likert scale from all investigators to a questionnaire on the easiness of use of spirometry and CAPTURE tool and its implementation in clinical practice once each center's inclusions had been completed.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier du Havre, Le Havre, Normandy, France